CLINICAL TRIAL: NCT06979141
Title: Comparative Study Between Efficacy of Dexmedetomidine, Magnesium Sulphate and Lidocaine for Cough Suppression During General Anesthetic Emergence
Brief Title: Dexmedetomidine, Magnesium Sulphate and Lidocaine for Cough Suppression After General Anesthesia
Acronym: MgSO4/DEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Talaat Abd Elhafeez Ahmed, Specialist. Mcs, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD/AZ.AST./AIP029/7/240/2/2025
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Dexmedetomidine; Magnesium Sulfate; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dexmedetomidine group ( D group ) (Active Comparator): Patients will receive 0.5 μg/kg dexmedetomidine in 10 ml normal saline 10 min before the end of surgery.
  Interventions: Drug: Dexmedetomidine
- Magnesium sulfate group ( M group ) (Active Comparator): Patients will receive 30 mg/kg IV magnesium sulfate 50% in 10 ml normal saline 10 min before the end of surgery.
  Interventions: Drug: Magnesium sulfate
- Lidocaine group ( L group ) (Active Comparator): Patients will receive lidocaine 1.5 mg/kg lidocaine in 10 ml normal saline 10 min before the end of surgery.
  Interventions: Drug: Lidocaine
- Control group ( C group ) (Placebo Comparator): Patients will receive 10 ml normal saline 10 min before the end of surgery.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive 0.5 μg/kg dexmedetomidine in 10ml normal saline 10 min before the end of surgery.
  Other Names: dex
  Arms: Dexmedetomidine group ( D group )
Drug: Magnesium sulfate — Patients will receive 30 mg/kg IV magnesium sulfate 50% 10 min before the end of surgery.
  Other Names: MgSO4
  Arms: Magnesium sulfate group ( M group )
Drug: Lidocaine — Patients will receive lidocaine 1.5 mg/kg lidocaine 10 min before the end of surgery.
  Arms: Lidocaine group ( L group )
Drug: normal saline — Patients will receive 10 ml normal saline 10 min before the end of surgery.
  Arms: Control group ( C group )

SUMMARY:
The aim of this prospective randomized controlled double-blinded study is to compare the efficacy of dexmedetomidine, MgSO4 and lidocaine for cough suppression during general anesthetic emergence as regard number and severity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-60 years.
* Both genders.
* Body mass index < 30 kg/ m2
* American Society of Anesthesiology (ASA) physical status I-II.
* Mallampati score class I or II.
* Patients undergoing surgery under general anesthesia.

Exclusion Criteria:

* Known allergy to study drugs.
* History of psychiatric illness.
* Patients with major organ diseases.
* Pre-existing neurological deficits.
* Body mass index >30 kg/m2.
* Active airway infection or history of tracheal and laryngeal surgery.
* Lower esophageal sphincter incompetence (and reflux).
* Increased intracranial and intraocular pressure.
* Use of cough-inducing medications
* Pregnant, and lactating women.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Cough suppression as regard number and severity. | at 0 and 10,20,30,40 minutes after endotracheal extubation.
  Coughing severity will be classified using the 3 point scale described by Minogue et al.: 1 = mild, single cough, 2 = moderate (lasting for <5 seconds) cough, and severe (lasting for >5 seconds) cough.

SECONDARY OUTCOMES:
Intraoperative heart rate (HR). | at 15-minutes interval.
  Changes in Intraoperative heart rate. change in heart rate per minute (HR/minute) will be all measured from the patient's arrival at the operating room to the end of surgery.
Intraoperative mean arterial blood pressure (MAP). | at 15-minutes interval.
  Changes in Intraoperative mean arterial blood pressure (MAP). change in mean arterial blood pressure (MAP) in mmHg will be all measured from the patient's arrival at the operating room to the end of surgery.
Intraoperative arterial oxygen saturation (Spo2). | at 15-minutes interval.
  Changes in Intraoperative arterial oxygen saturation (Spo2%). change in arterial oxygen saturation (Spo2%). be all measured from the patient's arrival at the operating room to the end of surgery.
Sedation score. | at 0,10,20,30, and 40 minutes after tracheal extubation.
  Sedation score will be recorded using the Ramsay sedation score (Ramsay et al., 1974).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud T Abd Elhafeez, Specialist.Mcs, Principal Investigator — mahmoud.talaat750@gmail.com
Locations (1):
- Faculty of Medicine, Al-Azhar university Assiut, Egypt., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No